



## **Prospective Clinical Study Protocol**

- Study to verify effectiveness and safety of at-home gait rehabilitation using wearable exoskeletal robot to improve gait in stroke patients, Investigator Initiated, Single center, Single group trial -

2024.08.05

[Severance Hospital]



## **Prospective Clinical Study Protocol**

#### 1. Title, stage, protocol identification number, revision history, etc.

- Title: Study to verify effectiveness and safety of at-home gait rehabilitation using wearable exoskeletal robot to improve gait in stroke patients, Investigator Initiated, Single center, Single group trial
- Stage: phase 4

#### 2. Summary of study plan

| Study objective | To evaluate the feasibility of a home-based robotic-assisted gait rehabilitation |
|---|---|
| | service using wearable exoskeletal robot for stroke patients |
| Study design overview | Investigator-initiated exploratory clinical study |
| | 4 weeks, pilot study |
| Drugs/medical devices for | Wearable exoskeletal robot |
| clinical trials | |
| Target number of subjects | Sixteen patients diagnosed with stroke |
| and calculation basis | This study aims to provide robotic-assisted gait training using wearable |
| | exoskeletal robot either at home or in nearby indoor spaces. The target number |
| | of participants was set based on clinical conditions. |
| | Rationale: The target number of participants was determined to be 16, considering |
| | a recruitment goal of two participants per month from among the outpatients at |
| | Yongin Severance Hospital, while accounting for dropout rates and clinical |
| | conditions. |
| Inclusion and exclusion | 1. Inclusion criteria |
| criteria | 1) adults aged 19 to 79 years (based on the age on their national ID at the time |
| | of consent) |
| | 2) individuals diagnosed with cerebral infarction or intracerebral hemorrhage |
| | confirmed by MRI or CT. |
| | 3) patients who have passed at least one month since stroke diagnosis. |
| | 4) individuals exhibiting spastic hemiplegic gait patterns due to stroke. |
| | 5) patients with a Functional Ambulatory Category score of less than 4. |
| | 6) individuals who can sit on the edge of a bed without assistance and stand for |



10 seconds with or without assistance.

- 7) individuals with sufficient cognitive ability to follow simple instructions and understand the study's content and purpose (Mini-Mental State Examination score >= 20)
- 2. Exclusion criteria
- 1) individuals with severe joint contractures or osteoporosis, or untreated fractures that contraindicate weight-bearing on the lower limbs.
- 2) individuals with skin conditions or open wounds that prevent device usage.
- 3) individuals with significant differences in leg length.
- 4) individuals with severe deformities or joint contractures in the lower limbs.
- 5) individuals at high risk of fractures due to conditions like osteoporosis.
- 6) individuals unable to maintain a sitting or standing position independently.
- 7) individuals with severe lower limb spasticity (Modified Ashworth Scale grade 2 or higher).
- 8) individuals with severe cognitive impairment (Mini-Mental State Examination score < 20), delirium, or severe language impairment that hinders cooperation with wearable exoskeletal robot gait training.
- 9) individuals unable to maintain prolonged standing or walking due to conditions like orthostatic hypotension or cardiopulmonary impairment.
- 10) individuals with conditions affecting gait, such as peripheral neuropathy, Parkinsonism, or those with alcohol dependence or severe diabetes.
- 11) pregnant women or those who could become pregnant.
- 12) individuals participating in other clinical trials.
- 13) individuals at high risk of falls or bleeding due to conditions like coagulopathies.
- 14) individuals shorter than 140 cm, taller than 190 cm, or weighing over 80 kg.
- 15) individuals with other clinical findings deemed inappropriate for the study by the principal investigator or study coordinator.

#### Study Methods

After obtaining informed consent, a screening test is conducted. The screening test includes a review of the participant's baseline symptoms and signs, medical history, and medication usage, followed by a physical examination and assessment of gait status, including the use of assistive devices and gait patterns. Participants who pass the screening test undergo an initial assessment within seven days.



The initial assessment includes physical function tests such as the 10-meter walk test, the Timed Up and Go (TUG) test, and the Berg Balance Scale, along with quality of life and Beck Depression Inventory assessments. Participants who complete the initial assessment begin robotic-assisted gait training within two days.

The training is conducted using a wearable exoskeletal robot for gait training at home or in nearby indoor spaces. The training lasts for four weeks, with sessions held 2-3 times per week, totaling 10 sessions, each lasting 30 minutes.

After four weeks, the robotic-assisted gait training concludes, and within two days, an endpoint assessment identical to the initial assessment is performed. Satisfaction with the wearable exoskeletal robot is also evaluated.

Any device malfunctions are addressed and documented. The usage and satisfaction levels of the wearable exoskeletal robot are analyzed, and pre- and post-training assessment metrics are compared.

#### Evaluation variable

- 1. Primary outcome measure
- Walking speed in the 10-meter walk test
- 2. Secondary outcome measures
- body composition analysis results
- spatiotemporal parameters of gait
- Timed Up and Go Test (TUGT)
- Berg Balance Scale (BBS)
- Satisfaction survey related to the use of the wearable exoskeletal robot based on the 12-item, 5-point K-QUEST scale

## Data analysis and statistical methods

1) Primary and secondary outcome measures

As a preliminary study exploring the efficacy and safety of home-based robotic-assisted gait training, the primary outcome measure is the walking speed in the 10-meter walk test before and after the intervention. The efficacy of the intervention will be evaluated by comparing pre- and post-intervention results using the Wilcoxon signed-rank test, with a p-value less than 0.05 indicating a significant difference due to the intervention.



Secondary outcome measures include quality of life scale, depression scale, body composition results, spatiotemporal gait parameters, Timed Up and Go Test, and Berg Balance Scale. These will also be compared pre- and post-intervention using the Wilcoxon signed-rank test, with statistical significance set at a p-value less than 0.05.

#### 2. Satisfaction evaluation

Satisfaction with the home-based robotic-assisted gait training will be analyzed using descriptive statistics to determine the mean, standard deviation, minimum, and maximum values for each item. Items with a mean score of 4 or higher will be interpreted as positive, while items with a mean score of 2 or lower will be interpreted as negative.

#### 3. Study background and theoretical basis

Out of the 2.6 million registered disabled individuals in Korea, 1.45 million are registered with physical and brain disabilities, accounting for 55% of the total registered disabilities (Source: Statistics Korea, 2020). Various causes such as stroke, cerebral palsy, spinal cord injury, and muscular dystrophy lead to functional impairments in the upper and lower limbs. According to a 10-year follow-up study on long-term functional levels in stroke rehabilitation, 48.3% of patients showed moderate to severe motor function decline at 6 months post-stroke, and 43.6% at 12 months, indicating a high demand for improving lower limb function and gait disabilities. Gait plays a crucial role in healthy skeletal and muscular development, improving cardiopulmonary function, 1-3 and performing daily activities, making the acquisition of walking ability a primary goal in rehabilitation therapy.

Various methods for gait rehabilitation training have been proposed,<sup>4</sup> with robotic-assisted gait training recently gaining attention. Continuous and repetitive training is essential for functional recovery following central nervous system injuries,<sup>5,6</sup> as it induces and enhances neuroplasticity. Robotic-assisted gait training facilitates accurate and repetitive walking patterns close to normal gait, overcoming discrepancies due to the therapist's experience, knowledge, and physical capabilities. Reports have shown that robotic-assisted gait training improves lower limb strength, gait and balance abilities, reduces depression, and enhances quality of life.<sup>7</sup> Various forms of gait-assistive robots are being attempted in clinical settings. Wearable gait-assistive robots,<sup>5</sup> compared to treadmill-based robots, offer precise and active training similar to actual walking, maximizing training effects. They are relatively compact, easily portable, and adjustable to individual patient characteristics.



The COVID-19 pandemic has increased the demand for healthcare services at home as well as within medical institutions. Despite significant advancements in rehabilitation robots due to developments in sensors, materials, near-field communication, and mobile applications, their use has been limited to medical institutions. This study aims to explore the feasibility of providing a home-based gait rehabilitation service using a wearable exoskeletal robot.

#### 4. Purpose of the study

Through pre- and post-intervention assessments, the study aims to determine the effectiveness of home-visit rehabilitation gait training using a wearable exoskeletal robot, conducted by a rehabilitation therapist under a doctor's diagnosis and prescription. This intervention consists of 10 sessions over four weeks, aiming to improve the gait function of stroke patients. Additionally, the study will evaluate the effectiveness and safety of home-based rehabilitation services by assessing patient satisfaction with the robotic-assisted gait training and conducting physical examinations post-intervention.

#### 5. Risk/benefit analysis

The study will use the Timed Up and Go Test (TUGT) to assess gait ability. This test is widely used in clinical settings and has a very low medical risk. To minimize the risk of falls during the test, participants will undergo sufficient practice under the supervision of the examiner before conducting the test in an environment equipped with safety bars.

Participants in this study will receive information about their muscle mass, gait, and balance abilities, and will benefit from systematic robotic-assisted gait training at home. The accumulated data during the study will be used to improve and enhance gait rehabilitation devices and to develop home-based services. Additionally, this data will contribute to research related to disease treatment and prognosis, thereby advancing medical knowledge and improving the quality of care. Therefore, the benefits gained from this study are expected to outweigh the potential risks.



#### 6. Target number of subjects and calculation basis

This study will be conducted on all patients visiting Yongin Severance Hospital who consent to participate and meet the selection criteria. The goal is to recruit two participants per month from the hospital's outpatients, with a target number of 10 participants, considering dropout rates and clinical conditions.

#### 7. Subject Inclusion/exclusion criteria

- 1) Inclusion criteria
- (1) adults aged 19 to 79 years (based on the age on their national ID at the time of consent)
- (2) individuals diagnosed with cerebral infarction or intracerebral hemorrhage confirmed by MRI or CT.
- (3) patients who have passed at least one month since stroke diagnosis.
- (4) individuals exhibiting spastic hemiplegic gait patterns due to stroke.
- (5) patients with a Functional Ambulatory Category score of less than 4.
- (6) individuals who can sit on the edge of a bed without assistance and stand for 10 seconds with or without assistance.
- (7) individuals with sufficient cognitive ability to follow simple instructions and understand the study's content and purpose (Mini-Mental State Examination score >= 20)
- 2) Exclusion criteria
- (1) individuals with severe joint contractures or osteoporosis, or untreated fractures that contraindicate weight-bearing on the lower limbs.
- (2) individuals with skin conditions or open wounds that prevent device usage.
- (3) individuals with significant differences in leg length.
- (4) individuals with severe deformities or joint contractures in the lower limbs.
- (5) individuals at high risk of fractures due to conditions like osteoporosis.
- (6) individuals unable to maintain a sitting or standing position independently.
- (7) individuals with severe lower limb spasticity (Modified Ashworth Scale grade 2 or higher).
- (8) individuals with severe cognitive impairment (Mini-Mental State Examination score < 20), delirium, or severe language impairment that hinders cooperation with wearable exoskeletal robot gait training.



(9) individuals unable to maintain prolonged standing or walking due to conditions like orthostatic hypotension or cardiopulmonary impairment.

(10) individuals with conditions affecting gait, such as peripheral neuropathy, Parkinsonism, or those with alcohol dependence or severe diabetes.

- (11) pregnant women or those who could become pregnant.
- (12) individuals participating in other clinical trials.
- (13) individuals at high risk of falls or bleeding due to conditions like coagulopathies.
- (14) individuals shorter than 140 cm, taller than 190 cm, or weighing over 80 kg.
- (15) individuals with other clinical findings deemed inappropriate for the study by the principal investigator or study coordinator.

#### 8. Information and management of clinical investigational drugs/medical devices

This study does not involve clinical trials; however, the following information and management methods pertain to the medical devices used in this study.

1) Wearable exoskeletal robot

(1) Item name: Wearable exoskeletal robot

(2) Classification number: A67080.01

(3) Packaging unit: 1 set

(4) Medical device class: Class III

(5) Model name: M20-A-C3, M20-B-C3

(6) Manufacturer: Angel Robotics Co., Ltd.

(7) Approval number: No. 22-857

(8) Appearance 엔젤렉스 M20-C

(9) Intended use: A robotic automation system used for muscle reconstruction and joint movement recovery







(10) Mechanism, usage, and precautions: Refer to the attached document

2) Device management

The wearable exoskeletal robot used in this study will be provided as one unit along with a robot transport cart

and gait aid tools, managed as follows:

(1) Security

The medical device used in this study will be stored according to the specified storage environment conditions in

a designated location (Spring County Jai Banquet Hall storage room) equipped with a locking mechanism.

Cooperation has been obtained from the institution's responsible person for the use of this location and locking

mechanism, and the medical device manager is responsible for security checks. (Refer to the attached document)

(2) Infection control

The medical device manager will conduct thorough disinfection procedures between sessions to minimize the risk

of cross-infection between participants. Before using the equipment, the manager will supervise the personal

hygiene of participants using hand sanitizers available in the indoor space where the gait training is conducted.

(3) Device transport and retrieval

The robotic-assisted orthopedic exercise device used in the study will be transported and retrieved using a robot

transport cart between the banquet hall where the gait training is conducted and the storage room where the

device is kept. These areas are connected spaces.

9. Study design (test group-control group, allocation, blinding and flow chart, etc.)

1) Study design overview

This investigator-initiated exploratory study will be conducted over a period of four weeks.

2) Experimental group

This study will include a single test group with a total of 10 participants. The selection of participants and the

entire treatment process using the wearable skeletal robot will be conducted according to the prescription and

guidance of a specialist in rehabilitation medicine, under the supervision of two occupational therapists. Participants

will receive robotic-assisted gait training twice a week for 30 minutes over four weeks, either at home or in nearby



indoor spaces such as a gym.

#### 3) Randomization and control group

This preliminary study follows a single-group design without randomization or a control group.

#### 4) Flowchart



#### 10. Study Methods

#### 1) Screening methods

The screening evaluation will be conducted by a specialist in rehabilitation medicine in an independent space, such as a consultation room, at Yongin Severance Hospital. After providing a thorough explanation of the study to the participants and obtaining their consent, the following steps will be taken:

- (1) Vital signs
- The examiner checks the participant's blood pressure, pulse, and temperature.
- (2) Physical examination



- 1 Manual muscle testing (lower limbs)
- The examiner evaluates the participant's lower limb manual muscle strength and joint range of motion according to the table below. The evaluation should be performed with the participant lying down or in a prone position, and the examiner can assist in changing positions if necessary.

| Score | Description |
|---|---|
| 0 | No palpable or observable muscle contraction |
| 1 | Palpable or observable contraction, but no motion |
| 1+ | Moves limb without gravity loading less than one half available $ROM^b$ |
| 2- | Moves without gravity loading more than one half ROMb |
| 2 | Moves without gravity loading over the full ROM <sup>b</sup> |
| 2+ | Moves against gravity less than one-half ROM <sup>b</sup> |
| 3- | Moves against gravity greater than one-half ROMb |
| 3 | Moves against gravity less over the full ROM <sup>b</sup> |
| 3+ | Moves against gravity and moderate resistance less than one-half ${\rm ROM}^b$ |
| 4- | Moves against gravity and moderate resistance<br>more than one-half $ROM^b$ |
| 4 | Moves against gravity and moderate resistance over the full $ROM^b$ |
| 5 | Moves against gravity and maximal resistance over the full $ROM^b$ |

<sup>&</sup>lt;sup>b</sup>ROM = range of motion.

- 2) Joint range of motion assessment (lower limbs)8
- The examiner evaluates the participant's lower limb manual muscle strength and joint range of motion using the table below as a reference. The assessment should be performed with the participant in a lying down or prone position, and the examiner can assist with position changes if necessary.
- < Joint Range of Motion Assessment Guide >

| | Low | er Extrem | iity | | |
|-----|-----------|-----------|-----------|-----|-----|
| Rt. | | | | | Lt. |
| 125 | flexion | | flexion | 125 | |
| 10 | extension | | extension | 10 | |
| 45 | abduction | 111- | abduction | 45 | |
| 10 | adduction | Hip | adduction | 10 | |
| 45 | E/R | | E/R | 45 | |
| 45 | I/R | | I/R | 45 | |
| 140 | flexion | | flexion | 140 | |
| 0 | extension | Knee | extension | 0 | |
| 20 | D/F | 4-17- | D/F | 20 | |
| 40 | P/F | Ankle | P/F | 40 | |

- 3 Spasticity assessment (Modified Ashworth Scale, MAS) (lower limbs)9
- The examiner evaluates the degree of spasticity in the participant's three major lower limb joints (hip, knee, ankle) to determine the extent of functional or stability impairment. The evaluation criteria are as follows:



| Score | |
|---|---|
| 0 | No increase in muscle tone |
| 1 | Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end range of motion when the part is moved |
| 1+ | Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range |
| 2 | More marked increase in muscle tone throughout most of the range, but affected part is easily moved |
| 3 | Considerable increase in muscle tone, passive movement is difficult |
| 4 | Affected part is rigid |

#### < Joint Spasticity Assessment Guide >

| Joint | Muscle | Right | Left | Joint | Muscle | Right | Left |
|---|---|---|---|---|---|---|---|
| | Flexors | | | Knee | Flexors | | |
| | Extensors | | | | Extensors | | |
| Hip | Abductors | | | Ankle | Dorsi-flexors | | |
| | Adductors | | | | Plantar-flexors | | |
| | Int. rotators | | | Foot | Invertors | | |
| | Ext. rotators | | | | Evertors | | |

- 4 Functional Ambulation Category (FAC)<sup>10</sup>
- The examiner evaluates the participant's postural stability during walking by observing and recording their gait according to the criteria below.

| Definition |
|------------------------------------------------------------------------------|
| Absolute inability to walk even with external help. |
| Requires external help to be able to walk. |
| Only able to walk on flat surfaces and known spaces like home. |
| Able to walk inside and outside of home but limited distances. |
| Able to walk anywhere but with obvious limp or need of technical assistance. |
| Normal deambulation. |

- ⑤ Mini-Mental State Examination (MMSE)<sup>11</sup>
- A standardized tool used to evaluate cognitive function and screen for dementia in a short period. The examiner asks the participant questions from the questionnaire and records the score based on the responses.



| Patient's Name: | Date: |
|-----------------|-------|
|-----------------|-------|

Instructions: Score one point for each correct response within each question or activity.

| Maximum<br>Score | Patient's<br>Score | Questions |
|---|---|---|
| 5 | | "What is the year? Season? Date? Day? Month?" |
| 5 | | "Where are we now? State? County? Town/city? Hospital? Floor?" |
| 3 | | The examiner names three unrelated objects clearly and slowly, then the instructor asks the patient to name all three of them. The patient's response is used for scoring. The examiner repeats them until patient learns all of them, if possible. |
| 5 | | "I would like you to count backward from 100 by sevens." (93, 86, 79, 72, 65,) Alternative: "Spell WORLD backwards." (D-L-R-O-W) |
| 3 | | "Earlier I told you the names of three things. Can you tell me what those were?" |
| 2 | | Show the patient two simple objects, such as a wristwatch and a pencil and ask the patient to name them. |
| 1 | | "Repeat the phrase: 'No ifs, ands, or buts."" |
| 3 | | "Take the paper in your right hand, fold it in half, and put it on the floor." (The examiner gives the patient a piece of blank paper.) |
| 1 | | "Please read this and do what it says." (Written instruction is "Close your eyes.") |
| 1 | | "Make up and write a sentence about anything." (This sentence must contain a noun and a verb.) |
| 1 | | "Please copy this picture." (The examiner gives the patient a blank piece of paper and asks him/her to draw the symbol below. All 10 angles must be present and two must intersect.) |
| 30 | | TOTAL |

#### (3) Bone Density Test<sup>12</sup>

The examiner evaluates the patient's risk of osteoporosis based on their medical history and current medications. If the patient is suspected to be at risk for osteoporosis but has not undergone testing in the past two years, a bone density test using dual-energy X-ray absorptiometry (DEXA) will be performed. Osteoporosis is diagnosed when the bone density of the spine or hip has a T-score of less than -2.5.<sup>13</sup>

#### (4) Pregnancy Test

The examiner assesses the patient's potential for pregnancy through medical history and measurement of chorionic gonadotropin hormone levels in urine.<sup>14</sup>

#### 2) Pre- and post-intervention evaluation variables

Before and after the intervention program, the research team will conduct the following tests or surveys on



participants in an independent space at Yongin Severance Hospital. The final evaluation will be conducted within 2 days after the intervention ends.

#### (1) Primary outcome measure

#### 1) 10MWT (10 meter walk test)

A simple and effective clinical evaluation method used to measure the walking speed of participants, useful for assessing functional recovery and changes in gait ability. The measurement method involves timing how long it takes to walk 10 meters, then dividing 10 by the time taken to record the walking speed (m/s).



#### (2) Secondary outcome measures

① Health-related quality of life measurement (36-item Short Form Survey Instrument, SF-36)

A self-reported survey consisting of 36 items used to assess participants' overall health-related quality of life. The evaluation tool measures satisfaction with overall health, with scores ranging from 0 to 100.15

| 36-ITEM SHORT FORM SI<br>INSTRUMENT (SF-36) | URVE | 1 | | INSTRUCTIONS During the past 4 weeks, have you had any of the following problems will daily activities as a result of your physical health? | th your work o | or other regular | INSTRUCTIONS These questions are about how your For each question, please give the or How much of the time during the part | ne ansv | wer that co | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient Name: | | | | | Yes | No | | All of | | | | | |
| Date of birth: | | | | 13. Cut down the <b>amount of time</b> you spent on work or other activities | 1 | 2 | | the | | A good bit<br>of the time | | e A little of<br>the time | None of the<br>time |
| INSTRUCTIONS Choose one option for each questionnaire item, | | | | 14. Accomplished less than you would like | 1 | 2 | 23. Did you feel full of pep? | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | 15. Were limited in the <b>kind</b> of work or other activities | 1 | 2 | 24. Have you been a very nervous | 1 | 2 | 3 | 4 | 5 | 6 |
| 1 - IN GENERAL, WOULD YOU SAY YOUR HEALTH IS: | | | _ | <ol> <li>Had difficulty performing the work or other activities (for example,<br/>it took extra effort)</li> </ol> | 1 | 2 | person<br>25. Have you felt so down in the | | 6 | | | | |
| 1 - Excellent 2 - Very good 3 - Go | _ | 4 - Fair | 5 - Poor | | | | dumps that nothing could cheer | 1 | 2 | 3 | 4 | 5 | 6 |
| 2 - COMPARED TO ONE YEAR AGO, HOW WOULD YOU RATE YOUR HEALTH IN GENERAL NOW? 1 - Much better now than a year ago | | | N GENERAL NOW? | INSTRUCTIONS | | | 26. Have you felt calm and peaceful? | 1 | 2 | 3 | 4 | 5 | 6 |
| 2 - Somewhat better now than a year ago<br>3 - About the same | | | | During the past 4 weeks, have you had any of the following problems with your work or other regular daily activities as a result of any emotional problems (such as feeling depressed or anxious)? | | | 27. Did you have a lot of energy? | 1 | 2 | 3 | 4 | 5 | 6 |
| 4 - Somewhat worse now than one year ago 5 - Much worse now than one year ago | | | | | Yes | No | 28. Have you felt downhearted and blue? | 1 | 2 | 3 | 4 | 5 | 6 |
| | | | | 17. Cut down the amount of time you spent on work or other activities: | 1 | 2 | 29. Did you feel worn out? | 1 | 2 | 3 | 4 | 5 | 6 |
| | NSTRUCTIONS he following Items are about activities you might do during a typical day. Does your health now limit ou in these activities? If so, how much? Circle the appropriate number. | | | 18. Accomplished less than you would like | 1 | 2 | 30. Have you been a happy person? | 1 | 2 | 3 | 4 | 5 | 6 |
| | los esta | | | 19. Didn't do work or other activities as carefully as usual | 1 | 2 | 31. Did you feel tired? | 1 | 2 | 3 | 4 | 5 | 6 |
| | Yes, limited<br>a lot | Yes, limited a | No, not limited at all | | | | | | | | | | |
| <ol> <li>Vigorous activities, such as running, lifting heavy<br/>objects, participating in strenuous sports</li> </ol> | 1 | 2 | 3 | 20. DURING THE PAST 4 WEEKS, TO WHAT EXTENT HAS YOUR PH | /SICAL HEAL | TH OR | 32. DURING THE PAST 4 WEEKS,<br>EMOTIONAL PROBLEMS INTERFE | | | | | | |
| Moderate activities, such as moving a table, pushing a vacuum cleaner, bowling, or playing golf | 1 | 2 | 3 | EMOTIONAL PROBLEMS INTERFERED WITH YOUR NORMAL SOCIA | | | FRIENDS, RELATIVES, ETC.)? | | | N SOCIAL P | | (Line visit | |
| Lifting or carrying groceries | 1 | 2 | 3 | FRIENDS, NEIGHBORS, OR GROUPS? | | | 1 - All of the 2 - Most of | the [ | 3 - Som | ne of the | 4 - A little | of5 - | - None of the |
| 6. Climbing several flights of stairs | 1 | 2 | 3 | 1 - Not at all 2 - Slightly 3 - Moderately 4 - Qu | ite a bit | 5 - Extremely | time time | | time | | the time | tin | 10 |
| 7. Climbing one flight of stairs | 1 | 2 | 3 | | | | INSTRUCTIONS How TRUE or FALSE is each of the form | ollowin | ig stateme | ents for you. | | | |
| 8. Bending, kneeling, or stooping | 1 | 2 | 3 | 21. HOW MUCH BODILY PAIN HAVE YOU HAD DURING THE PAST 4 | WEEKS? | | | 1 | Definitely | | | | Definitely |
| 9. Walking more than a mile | 1 | 2 | 3 | 1 - None 2 - Very mild 3 - Mild 4 - Moderate 5 | - Severe | 6 - Very severe | | | true | Mostly true | Don't know | w Mostly fals | false |
| 10. Walking several blocks | 1 | 2 | 3 | | | | <ol> <li>I seem to get sick a little easier<br/>other people</li> </ol> | than | 1 | 2 | 3 | 4 | 5 |
| 11. Walking one block | 1. | 2 | 3 | 22. DURING THE PAST 4 WEEKS, HOW MUCH DID PAIN INTERFERE | WITH YOUR | NORMAL | 34. I am as healthy as anybody I kno | w | 1 | 2 | 3 | 4 | 5 |
| 12. Bathing or dressing yourself | 1 | 2 | 3 | WORK (INCLUDING BOTH WORK OUTSIDE THE HOME AND HOUSE | WORK)? | | 35. I expect my health to get worse | | 1 | 2 | 3 | 4 | 5 |
| | | | | 1 - Not at all 2 - A little bit 3 - Moderately 4 - Q | ite a bit | 5 - Extremely | 36. My health is excellent | | 1 | 2 | 3 | 4 | 5 |

#### 2 Beck depression inventory (BDI)<sup>16</sup>

An evaluation tool designed based on clinical depressive symptoms. It consists of 21 self-reported items where



patients check and record their scores in areas such as affective cognition and motivation. Scores range from 0 to 63.



#### 3 Body composition analysis

This is a test performed to check the subject's limb muscle mass, and the test method is as follows.

- Perform body composition analysis<sup>17</sup> based on bioimpedance analysis.
- To ensure accurate measurement, the test subject is instructed to empty his/her bladder before the test and not to consume caffeinated beverages, eat, drink, or perform strenuous exercise for one hour prior to the test.
- To correct for muscle mass differences due to height, use the calculated value of limb muscle mass (Appendicular skeletal mass) divided by the square of the height.







#### 4 Spatiotemporal parameters of walking

Spatiotemporal parametric data of gait collected while the subject is performing a home-based activity wearing an insole gait analyzer, recording total steps, steps per minute, gait speed (km/h), distance walked (m), stride length (m), and swing phase rate (%).

- Step count: The number of steps measured while walking.
- Cadence: The number of steps taken per minute, with the unit being steps/min (spm). Normal values are  $\geq 70$  steps/min for those under 65 years old and  $\geq 60$  steps/min for those 65 years and older.
- Gait speed: The speed of walking, with the unit being km/h. Normal values are  $\geq$  2.0 km/h for those under 65 years old and  $\geq$  1.5 km/h for those 65 years and older.
- Distance: The total distance traveled while walking, measured in meters (m).
- Stride length: The distance from the heel of one foot to the heel of the same foot in the next step. The distance is measured in meters (m), and it is normalized for height by dividing stride length by height. Normal values are  $\geq$  0.5 m/height for those under 65 years old and  $\geq$  0.4 m/height for those 65 years and older.
- Swing ratio: The percentage of the gait cycle that is in the swing phase, with the unit being %. Normal values are  $\geq$  30% for those under 65 years old and  $\geq$  28% for those 65 years and older.

#### (5) Timed up and go test (TUG)

The above test assesses walking speed along with balance ability during walking <sup>18</sup>, and this is performed as follows.

- A 46 cm high armrest chair, a color cone is placed at a distance of 3 meters from the chair and the subject is instructed to sit on the chair.
- In the preparation phase, the subject leans against the chair backrest and places his/her arms on the armrests, then stands up on the instruction "Start", walks 3 meters, turns around the color cone, returns to the starting point and sits down on the chair.



#### 6 Berg Balance Scale

The following tests evaluate static and dynamic balance,<sup>19</sup> and have been used in previous studies to assess



progress after robotic-assisted gait therapy.<sup>20</sup> The examiner instructs the participant to perform the following 14 tasks and evaluates them according to specific criteria. Scores range from 0 to 56.

| Balance Section | | S | cor | e. | |
|-----------------------------------------|-----|---|-----|----|----|
| Sitting to standing | 0 | 1 | 2 | 3 | 4. |
| Standing unsupported | 0 | 1 | 2 | 3 | 4. |
| Sitting unsupported- | 0 | 1 | 2 | 3 | 4. |
| Standing to sitting | 0 | 1 | 2 | 3 | 4. |
| Transfers+ | 0 | 1 | 2 | 3 | 4. |
| Standing with eyes closed <sub>e</sub> | 0 | 1 | 2 | 3 | 4. |
| Standing with feet together | 0 | 1 | 2 | 3 | 4. |
| Reaching forward with outstretched arme | 0 | 1 | 2 | 3 | 4 |
| Retrieving object from floor | 0 | 1 | 2 | 3 | 4. |
| Turning to look behind↔ | 0 | 1 | 2 | 3 | 4. |
| Turning 360 degreese | 0 | 1 | 2 | 3 | 4. |
| Placing alternate foot on stool€ | 0 | 1 | 2 | 3 | 4. |
| Standing with one foot in front | 0 | 1 | 2 | 3 | 4. |
| Standing on one foot∘ | 0 | 1 | 2 | 3 | 4. |
| Total Sco | ore | | | / | 56 |

#### 3) Satisfaction evaluation

Participants will complete a satisfaction survey for the home-based rehabilitation service using the wearable exoskeletal robot, based on the Korean version of the Quebec User Evaluation of Satisfaction with assistive Technology (K-QUEST 2.0).<sup>21</sup> This survey consists of 12 items on a 5-point scale. Participants rate their satisfaction with the assistive device and related services as follows:

1: Very dissatisfied, 2: Dissatisfied, 3: Neutral, 4: Satisfied, 5: Very satisfied

Participants are instructed to provide reasons if they do not select "very satisfied" for any item.

| 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|



| Is it convenient to adjust (fix and lock) parts of the wearable exoskeletal robot? Reason: | | | |
|---|---|---|---|
| Do you think the wearable exoskeletal robot is safe and sturdy? Reason: | | | |
| Are you satisfied with the durability (long-term usability) of the wearable exoskeletal robot? Reason: | | | |
| Was the method of using the wearable exoskeletal robot convenient? Reason: | | | |
| Do you think the wearable exoskeletal robot is comfortable to wear? Reason: | | | |
| Are you satisfied with the effectiveness (purposeful use) of the wearable exoskeletal robot? Reason: | | | |
| Are you satisfied with the service and delivery program (delivery process, time required) of the wearable exoskeletal robot? Reason: | | | |
| Are you satisfied with the repair and maintenance service of the wearable exoskeletal robot? Reason: | | | |
| Are you satisfied with the professional services (information, precautions) provided while using the wearable exoskeletal robot? Reason: | | | |
| Are you satisfied with the after-sales service (continuous maintenance service) of the wearable exoskeletal robot? Reason: | | | |
| - Please mark the three items participants consider most important among the 12 | 2 satisfa | action | items. |

| | Ο 표시 |
|---------------------|------|
| 1. Specifications | |
| 2. Weight | |
| 3. Convenience | |
| 4. Safety | |
| 5. Durability | |
| 6. Usability | |
| 7. Comfort | |
| 8. Effectiveness | |
| 9. Service delivery | |



| 10. Repair and maintenance services |
|-------------------------------------|
| 11. Professional services |
| 12. After-sales service |

#### 4) Home-based robotic-assisted gait training

The participant's robotic-assisted gait training is conducted in collaboration with the research team (physical therapist or occupational therapist) under the prescription and guidance of a rehabilitation medicine specialist as follows. The gait training program begins within 2 days of the initial assessment and is conducted at home or in an indoor environment similar to the home setting. No transportation support, such as vehicles, is provided.

(1) Warm-up exercises before wearing the robot

Participants perform stretching exercises for 5 minutes before wearing the wearable exoskeletal robot.

#### (2) Application of the wearable exoskeletal robot

The wearable exoskeletal robot used in this study is a medical device that assists the hip and knee joints during gait training to achieve a near-normal walking trajectory. The evaluator applies this device to the participant and provides gait training on level ground. The robot can provide assistive torque during various walking phases, automatically detected through combined information from ground contact sensors, encoders (incremental and absolute) of the actuators, and inertial measurement unit sensors. According to the polynomial assistive joint torque profile by gait phase, flexion torque is generated in the hip and knee joints during the swing phase, and extension torque is generated in the hip and knee joints during the stance phase, aiding the participant's gait. The therapist aims to train the participant to walk in a pattern as close to normal as possible for the maximum duration. The gait training program consists of 10 sessions over 4 weeks, conducted 3 times a week for 30 minutes each session. All training sessions are conducted under the supervision of two research team members (physical therapists or occupational therapists). If the participant cannot continue the 30-minute session due to muscle endurance decline or pain, the gait training is terminated, and the actual session duration and the reasons for early termination are recorded.

#### (3) Recording adverse reactions and device malfunctions

- The research team (physical therapists or occupational therapists) records the types and frequencies of safety incidents and reasons for device malfunctions that occur during the participant's gait training.
- If adverse reactions such as pain occur, the type, severity, frequency, name of the adverse reaction, onset and resolution dates, characteristics, and causality are investigated and recorded.



5) Definition of analysis groups, missing data, and outlier management plan

#### (1) Definition of analysis groups

The analysis groups consist of all participants undergoing robotic-assisted gait training. The analysis includes their age, diagnosis, physical function assessments, and extracted gait parameter data.

#### (2) Missing data and outlier management plan

In cases of missing data due to study withdrawal or dropout, the Complete Case Analysis method is used, which analyzes only completely observed cases. Data from sessions with missing values are excluded from the analysis. Outliers identified using box plots and quartiles are also excluded from the analysis to maintain data integrity and enhance the study's accuracy and reliability. Information about the excluded participants is presented.

#### 6) Comparative analysis of pre- and post-intervention differences

After the completion of the gait training program using the wearable exoskeletal robot, the evaluator performs a comparative analysis of the collected data from participants following the final assessment and satisfaction survey.

#### 11. Study procedures and evaluation

| Phase | Screening / Initial assessment | Intervention | | | Final assessment |
|---|---|---|---|---|---|
| week | 0 | 1 | 2 | 3 | 4 |
| written consent | 0 | | | | |
| Inclusion/exclusion criteria | 0 | | | | |
| Demographic information and antecedent history | 0 | | | | |
| Primary outcome measure 10MWT (10 meter walk test) | 0 | | | | 0 |
| Secondary outcome measures | 0 | | | | 0 |



| Health-related quality of life measurement | | | | |
|--------------------------------------------|---|---|---|---|
| Beck depression inventory | | | | |
| Body composition analysis | | | | |
| Spatiotemporal parameters of | | | | |
| walking | | | | |
| Timed up and go test (TUG) | | | | |
| Berg Balance Scale | | | | |
| Satisfaction evaluation | | | | 0 |
| Home-based robotic-assisted gait training | 0 | 0 | 0 | 0 |

#### 12. Criteria for stopping and dropping out of the study

If a participant discontinues their participation in this clinical trial, only the information collected up to that point will be used in the study. The data will be stored for three years after the study ends and then destroyed.

1) Termination and early suspension

#### (1) Withdrawal of consent

If the participant or their legal representative withdraws consent before the end of the study, only the information collected up to that point will be used. The data will be stored for three years after the study ends and then destroyed.

(2) Occurrence of serious adverse events

#### 2) Dropout

If the participant's early discontinuation is not due to withdrawal, their willingness to continue providing information for the study will be reconfirmed. If they agree, the information collected up to the point of dropout will be anonymized and used in the study.



(1) The medical team determines that there is a serious medical necessity preventing the participant from continuing in the clinical study.

(2) The participant uses concurrent surgery, medications, or other medical devices that may affect the safety and

efficacy evaluations.

(3) The participant does not comply with the investigator's instructions or the terms of the consent form, affecting

the evaluation of efficacy.

(4) The participant's absence prevents continuous observation.

(5) Other cases where the principal investigator determines there are issues in continuing the clinical trial.

3) Handling of discontinuation and dropout

(1) If a participant drops out, the reason for dropout and the clinical trial-related data collected up to the point of

dropout will be recorded and stored.

(2) If a participant is unable to visit during the study, their status must be confirmed, and the reason for their

absence must be clearly documented.

(3) Participants who drop out without valid reasons or justification will be included in the statistical analysis for

efficacy and safety evaluation.

13. Safety evaluation criteria, evaluation methods, and reporting methods, including adverse

reactions

1) Evaluation criteria

To ensure the safety of study participants, the principal investigator will act as the safety monitor, conducting

monitoring and evaluating safety.

(1) Symptoms reported by participants or identified through physical examinations during or after the intervention

in the control and experimental groups (e.g., musculoskeletal pain and skin lesions during gait training).

(2) Physical examinations (e.g., musculoskeletal abnormalities and skin lesions such as erythema and edema at the

site of the wearable exoskeletal robot application).



- (3) Safety evaluation related to falls:
- Number of falls
- Severity of injuries caused by falls (e.g., bruises, fractures, other injuries)
- Other

#### 2) Evaluation method

- (1) Perform statistical analysis to evaluate the severity and type of adverse reactions and the incidence rates of adverse reactions in the experimental and control groups, based on reports from participants or physical examinations.
- (2) Safety analysis will be conducted with a significance level of <0.05 (two-sided).
- 3) Adverse event reporting
- (1) Reporting subjects: All participants in this clinical trial.
- (2) Adverse event evaluation criteria:
- Evaluate the cause of adverse events according to the following criteria:
- Device-related issues: Adverse events caused by device malfunction, breakdown, or damage despite following the intended use, method of use, and precautions specified by the manufacturer.
- Procedural issues: Adverse events caused by the procedure itself when the device was used correctly and there were no issues with the patient's condition or underlying disease.
- Patient-related issues: Adverse events caused by the patient's condition or underlying disease when the device was used correctly and the procedure was performed correctly.
- Evaluation impossible: When the adverse event report does not match the actual product or multiple causes are involved, making it impossible to determine the cause.
- (3) Adverse event evaluation method
- The clinical trial investigator will record symptoms, onset date, and resolution date of adverse reactions in an adverse reaction record form if an adverse reaction occurs during the trial.
- (4) Adverse event reporting method:
- This content will be reported according to the regulations related to medical device clinical trials and the standard operating procedures (SOPs) specified by the clinical trial institution and the institution's IRB regulations.



#### I. Definition of terms

- "Safety information" refers to data or information related to the safety and efficacy of approved, certified, or reported medical devices, including cases of adverse effects.
- "Adverse effect information" refers to cases of adverse effects or potential adverse effects occurring domestically or internationally during the handling or use of medical devices.
- "Side effect" refers to any unintended result, suspected to have occurred due to normal use of the medical device, including unintended desirable results.
- "Adverse event" refers to undesirable outcomes among side effects, not necessarily having a causal relationship with the medical device.
- "Serious adverse event" refers to an adverse event that meets any of the following criteria:
- a. Results in death or life-threatening adverse effects
- b. Requires hospitalization or prolongation of existing hospitalization
- c. Causes permanent or significant disability or incapacity
- d. Results in congenital anomalies or birth defects
- "Unexpected adverse event" refers to an adverse event that differs in severity, specificity, or outcome from what is described in the approved, certified, or reported information of the medical device.

#### II. Safety evaluation criteria

Safety evaluation criteria refer to the standards for recording the severity of anticipated adverse effects and adverse reactions in case report forms.

#### III. Safety evaluation methods

The methods for safety evaluation include statistical analysis techniques and evaluation criteria for comparative assessment of the frequency of occurrence of adverse effects, abnormal device responses, and adverse reactions associated with clinical trial medical devices.



IV. Reporting adverse reactions

- Serious adverse reactions at each institution must be reported to the clinical trial coordinator

and monitoring staff via email within 48 hours of awareness.

- The principal investigator must report serious adverse reactions to the institution's IRB

according to IRB regulations and provide additional detailed reports as specified in the

protocol.

- In cases of death or life-threatening situations, the principal investigator must report to the

head of the Food and Drug Administration within 7 days of becoming aware of the event. For

other serious and unexpected adverse reactions, the report must be submitted within 15 days.

4) Monitoring Plan for Participants Who Experience Adverse Events

(1) This is a preliminary case study with a low risk level, requiring minimal invasive intervention. Therefore, weekly

monitoring will be conducted under the supervision of the principal investigator. This monitoring will ensure data

completeness by cross-checking supporting documents, case report forms (CRF), and protocols, and reviewing

safety data of the study participants.

(2) Participants who experience adverse events will be compensated according to the provisions of the compensation

protocol in this study plan. Monitoring of the treatment progress will continue until the adverse reaction is resolved

or until the participant's scheduled study completion.

(3) For participants who experience adverse events and do not refuse follow-up, the progress of the adverse events

will be observed through reported symptoms and physical examinations at scheduled study visits.

5) As a preliminary case study with a low risk level requiring minimal invasive intervention, weekly monitoring will

be conducted under the supervision of the principal investigator. This will ensure data completeness by cross-

checking supporting documents, CRF, and protocols, and reviewing the safety data of study participants.

6) Participants in the study can decide to discontinue their participation at any time if they feel discomfort related

to the study. The principal investigator or study coordinator will fully explain and confirm this when obtaining

consent from participants.

7) In the event of any violations or deviations from the study, the situation and the researcher's actions and

preventive measures will be promptly reported to the IRB in writing. Immediate treatment and observation will be

provided if participants are injured or if new incidents occur during the evaluation, with a thorough investigation

of the causes. Treatment will follow the hospital's standard procedures. These incidents will be reported in interim

reports and included in the research paper. However, this study is considered to have a low likelihood of future

adverse effects, and therefore no additional treatment costs have been budgeted.

14. Data analysis and statistical considerations

1) Primary and secondary outcome measures

This study is a preliminary exploration of the efficacy and safety of home-based robotic-assisted gait training. The

primary evaluation variable is the walking speed measured by the 10-meter walk test before and after robotic-

assisted gait rehabilitation. The pre- and post-intervention results will be compared using the Wilcoxon signed-rank

test, with a p-value of less than 0.05 indicating a significant difference due to the intervention.

Secondary evaluation variables include quality of life scale, depression scale, body composition results,

spatiotemporal gait parameters, Timed Up and Go test, and Berg Balance Scale. These will also be compared pre-

and post-intervention using the Wilcoxon signed-rank test, with statistical significance set at a p-value of less than

0.05.

The results of the satisfaction with home-based robotic-assisted gait training will be analyzed using descriptive

statistics, identifying the mean, standard deviation, minimum, and maximum values for each item. Items with an

average score of 4 or higher will be interpreted as positive, while items with an average score of 2 or lower will be

interpreted as negative.

2) Satisfaction evaluation:

The satisfaction with the home-based gait rehabilitation service using the wearable exoskeletal robot will be

analyzed using descriptive statistics, presenting the mean, standard deviation, median, minimum, and maximum

values.

15. Measures to protect personal information and maintain confidentiality of study data

(A)

Severerance: M20\_20240805

1) Protection of the subject's identity

When seeking consent for study, the study is explained to the subject and consent is obtained in an independent

space in the counseling room within the outpatient department of the Rehabilitation Medicine Department.

All information collected from this study must be kept secret from anyone other than the researchers involved in

the study and it is used for study purposes only. Sensitive personal information that can identify individuals will not

be shared with organizations other than the hospital and will go through an anonymization process (deidentification).

Anonymization is achieved by using the unique number of the insole-type gait analyzer issued to the subject, and

data collected through the application will be stored in accordance with the medical device company's security

policy and will be discarded after the end of the study, and will be de-identified before being forwarded to the

medical device company. De-anonymization is limited to cases where it is necessary in relation to the individual's

treatment. Only the final results of the analysis are disclosed to medical device companies and ownership of the

data lies with the hospital.

2) Confidentiality of study materials

In the case of documentary data, it will be kept in a locked device to prevent it from being exposed to others,

stored on a computer with restricted access, and managed by the researcher in charge.

3) Preservation of records

Study-related data are stored for 3 years in accordance with the Enforcement Rules of the Bioethics Act (Human

subject researchers must keep records pursuant to Paragraph 1 for 3 years from the end of study), and among

documents that have expired the retention period, subject related personal information shall be destroyed in

accordance with Article 16 of the Enforcement Decree of the Personal Information Protection Act. However, if storage

of the data is necessary for follow-up study, record accumulation, etc., the retention period must be extended after

deliberation by the institutional committee.

16. Management, storage, and disposal measures when collecting human materials, genetic

information, etc.

No human specimens or genetic information are collected in this study.



#### 17. Subject recruitment method and consent procedure

After approval from the Yongin Severance Hospital IRB, among the visitors to Yongin Severance Hospital who decided and agreed to participate voluntarily in this study, interviews are conducted in an independent space, an explanatory statement approved by the IRB is provided, and consent forms are obtained.

After providing a sufficient explanation regarding participation in the clinical trial, the consent form must be completed in a non-oppressive environment, and when writing the consent form, participants must be explained that consent can be withdrawn at any time, so that they participate in the clinical trial. In addition, the intention to participate in the study is confirmed during the conduct of the study test, so that consent can be withdrawn at any time at the person's discretion.

#### 18. Protection measures when recruiting vulnerable subjects

This study does not recruit vulnerable subjects.

# 19. Information on the principal investigator and participating researchers, location of study conduct, and study period

#### (1) Principal investigator

| Name | Affiliated organization | Major | Job title | Phone |
|---|---|---|---|---|
| Na Young<br>Kim | Yonsei University College of Medicine Yongin Severance | Rehabilitation<br>medicine | Assistant<br>Professor | 031-5189-8163<br>Kny8452 @yuhs.ac |
| | Hospital | | | |

#### 2) Test manager

The test manager checks whether the test subject meets the selection criteria at the testing institution and manages the overall process of the experiment.



| Name | Affiliated organization | Major | Job title | Phone |
|---|---|---|---|---|
| Na Young<br>Kim | Yonsei University College of Medicine Yongin Severance Hospital | rehabilitation<br>medicine | Assistant<br>Professor | 031-5189-8163<br>Kny8452 @yuhs.ac |
| Seung Ick<br>Choi | Yonsei University<br>College of Medicine | Department<br>of Integrative<br>Medicine | Integrated<br>course<br>graduate<br>student | 010-8821-5297<br>rehab1@yuhs.ac |
| So Jeong<br>Lim | Yonsei University<br>Industry-Academic<br>Cooperation Foundation | occupational<br>therapy | researcher | 010-2971-3773<br>rehab2@yuhs.ac |
| Hwi Woo<br>Yang | Yonsei University Industry-Academic Cooperation Foundation | occupational<br>therapy | researcher | 010-7360-4439<br>rehab5@yuhs.ac |

#### 3) Medical device manager

| Name | Affiliated organization | Major | Phone |
|---|---|---|---|
| Seung Ick<br>Choi | Yonsei University<br>College of Medicine | Integrated<br>course<br>graduate<br>student | 010-8821-5297<br>rehab1@yuhs.ac |

### 20. Location and duration of study

#### 1) Location of study

| Organization name | Location | Phone |
|-------------------|----------|-------|



| Yonsei University | | |
|---------------------|------------------------------------|---------------|
| College of Medicine | 363 Dongbaekjukjeon-daero, | 031-5189-8891 |
| Yongin Severance | Giheung-gu, Yongin-si, Gyeonggi-do | |
| Hospital | | |

#### 2) Period

24 months after IRB approval

#### 21. Data safety monitoring plan

The safety inspector (principal investigator) monitors the overall study progress at monthly intervals to ensure the completeness of the data, including the status of the study, whether the registration subjects are suitable for the selection criteria, the appropriateness of the consent acquisition procedure, whether violations/deviations from the study plan have occurred, and whether the subjects have had adverse reactions.

#### 22. Study plan (schedule table)

| Detailed development | Detailed schedule (months) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| items | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
| Study protocols and IRB approval | | | | | | | | | | | | |
| Subject Recruitment | | | | | | | | | | | | |
| Conduct of study procedures and follow- up period | | | | | | | | | | | | |



| Detailed development | Detailed schedule (months) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| items | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 21 | 22 | 23 | 24 |
| Subject Recruitment | | | | | | | | | | | | |
| Conduct of study procedures and follow- up period | | | | | | | | | | | | |

#### 23. References

- 1. Salzman B. Gait and balance disorders in older adults. American family physician 2010;82:61-68
- 2. Bennett DA, Beckett LA, Murray AM, Shannon KM, Goetz CG, Pilgrim DM, et al. Prevalence of parkinsonian signs and associated mortality in a community population of older people. New England Journal of Medicine 1996;334:71-76
- 3. Lange AK, Vanwanseele B, Fiatarone singh MA. Strength training for treatment of osteoarthritis of the knee: a systematic review. Arthritis Care & Research: Official Journal of the American College of Rheumatology 2008;59:1488-1494
- 4. Chou C-H, Hwang C-L, Wu Y-T. Effect of exercise on physical function, daily living activities, and quality of life in the frail older adults: a meta-analysis. Archives of physical medicine and rehabilitation 2012;93:237-244
- 5. De Luca R, Maresca G, Balletta T, Cannavò A, Leonardi S, Latella D, et al. Does overground robotic gait training improve non-motor outcomes in patients with chronic stroke? Findings from a pilot study. Journal of Clinical Neuroscience 2020;81:240-245
- 6. Chin L, Lim W, Kong K. Evaluation of robotic-assisted locomotor training outcomes at a rehabilitation centre in Singapore. Singapore medical journal 2010;51:709
- 7. Schwartz I, Meiner Z. Robotic-assisted gait training in neurological patients: who may benefit? Annals of biomedical engineering 2015;43:1260-1269
- 8. Gajdosik RL, Bohannon RW. Clinical measurement of range of motion: review of goniometry emphasizing reliability and validity. Physical therapy 1987;67:1867-1872



- 9. Gregson JM, Leathley M, Moore AP, Sharma AK, Smith TL, Watkins CL. Reliability of the Tone Assessment Scale and the modified Ashworth scale as clinical tools for assessing poststroke spasticity. Archives of physical medicine and rehabilitation 1999;80:1013-1016
- 10. Mehrholz J, Wagner K, Rutte K, Meiβner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Archives of physical medicine and rehabilitation 2007;88:1314-1319
- 11. Tombaugh TN, McIntyre NJ. The mini-mental state examination: a comprehensive review. Journal of the American Geriatrics Society 1992;40:922-935
- 12. Plank LD. Dual-energy X-ray absorptiometry and body composition. Current Opinion in Clinical Nutrition & Metabolic Care 2005;8:305-309
- 13. Rachner TD, Khosla S, Hofbauer LC. Osteoporosis: now and the future. The Lancet 2011;377:1276-1287
- 14. Chard T. Pregnancy tests: a review. Human reproduction 1992;7:701-710
- 15. Anderson C, Laubscher S, Burns R. Validation of the Short Form 36 (SF-36) health survey questionnaire among stroke patients. Stroke 1996;27:1812-1816
- 16. Richter P, Werner J, Heerlein A, Kraus A, Sauer H. On the validity of the Beck Depression Inventory: A review. Psychopathology 1998;31:160-168
- 17. Andreoli A, Garaci F, Cafarelli FP, Guglielmi G. Body composition in clinical practice. European journal of radiology 2016;85:1461-1468
- 18. Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. Journal of chronic diseases 1987;40:373-383
- 19. Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Physical therapy 2013;93:158-167
- 20. Bang D-H, Shin W-S. Effects of robot-assisted gait training on spatiotemporal gait parameters and balance in patients with chronic stroke: A randomized controlled pilot trial. NeuroRehabilitation 2016;38:343-349
- 21. Lee S-H, Jung B-K, Park S-Y. Korean translation and psychometric properties of Quebec user evaluation of satisfaction assistive technology 2.0. Journal of the Korea Academia-Industrial Cooperation Society 2013;14:3284-3292
- 22. Nedergård H, Arumugam A, Sandlund M, Bråndal A, Häger CK. Effect of robotic-assisted gait training on



objective biomechanical measures of gait in persons post-stroke: a systematic review and meta-analysis. Journal of Neuroengineering and Rehabilitation 2021;18:1-22

23. Park G-M, Cho S-H, Hong J-T, Kim D-H, Shin J-C. Effects and safety of wearable exoskeleton for robot-assisted gait training: a retrospective preliminary study. Journal of personalized medicine 2023;13:676